CLINICAL TRIAL: NCT05872984
Title: The Evaluation of the Influence of the Use of Total Blood Volume Measurement During Dialysis on the Incidence of Intradialytic Hypotension Associated Events
Brief Title: Evaluation of Total Blood Volume Measurement During Dialysis on the Incidence of Intradialytic Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HagaZiekenhuis (Other)
Responsible Party: Principal Investigator, Louis Jean Vleming, dr. LJ Vleming, HagaZiekenhuis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL71892.058.19
Record Dates: First submitted 2023-04-25; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Hemodialysis Complication; Hypotension During Dialysis; Diagnostic Tests
Keywords: Hemodialysis; Intradialytic hypotension; Intradialytic morbid events

STUDY DESIGN:
Intervention Model Description: The intervention consists of the adjustment of the patients' dry weight, based on absolute blood volume measurement. Dry weight will be adjusted at the start of the intervention period in all subjects in the intervention group with a normalized blood volume below 65 ml/kg, regardless the occurrence of intradialytic hypotension associated adverse events during the baseline period. Dry weight will be increased once with 0,5kg.
Masking Description: Both the patients and the clinicians involved in patient care were not aware of the results of the absolute blood volume measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm: adjustment of dry weight based on absolute blood volume measurement (Experimental): Dry weight will be adjusted at the start of the intervention period in all subjects in the intervention group with a normalized blood volume below 65 ml/kg, regardless the occurrence of intradialytic hypotension associated adverse events during the baseline period. Dry weight will be adjusted once with 0,5kg.
  Interventions: Diagnostic Test: adjustment of dry weight based on absolute blood volume measurement
- Control arm: standard care (No Intervention): standard care provided by the clinician, no intervention.

INTERVENTIONS:
Diagnostic Test: adjustment of dry weight based on absolute blood volume measurement — adjustment of dry weight based on absolute blood volume measurement
  Arms: Intervention arm: adjustment of dry weight based on absolute blood volume measurement

SUMMARY:
Establishing the euvolemic state in hemodialysis patients -the so called "dry weight"- is an important clinical conundrum in every nephrologist's daily practice. Underestimation of dry weight (with excessive ultrafiltration) results in dialysis-induced hypotension. Currently used methods to establish dry weight, including clinical assessment, bio-impedance spectroscopy and online relative blood volume (RBV) measurements, all have their limitations. RBV measurement reflects changes in blood volume during dialysis without providing any information about the initial hydration status, or the initial absolute blood volume (ABV). Recently, researchers proposed a new method to calculate ABV, by using the principle of dilution-indicator with RBV measurement. In a small cohort study they identified a total blood volume threshold of 65 millilitres per kilogram dry weight predicting for intra-dialytic hypotension associated symptoms.

The goal of current clinical trial is to re-investigate the accuracy of the above-described method and to confirm the hypothesis of a critical threshold of 65 ml blood volume per kg dry weight in haemodialysis patients. Researchers will compare adjustment of dry weight based on the ABV measurement with standard care to see if dialysis-induced hypotension will be reduced.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patients of three dialysis locations of the Haga Hospital (Zoetermeer, The Hague Leyweg and The Hague Sportlaan).
* Maintenance hemodialysis, with initiation of treatment predates inclusion in the study by at least 3 months.
* Hemodialysis scheme three times weekly for four hours
* Age above 18 years.

Exclusion Criteria:

* Clinically relevant fistula dysfunction resulting in single poold Kt/V <1,2
* Severe volume overload with a contraindication to bolus fluid infusion during dialysis according to the treating physician.
* Severe cardiac dysfunction responsible for >1x intradialytic hypotension associated adverse event /week according to treating physician
* Severe liver failure with or without presence of ascites
* More than three hemodialysis sessions per week
* Single needle treatment
* Central venous access
* Residual diuresis > 500 ml/ 24h
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
difference in the incidence of intradialytic hypotension-associated adverse events between the intervention and control group | 10 weeks
  The incidence of intradialytic hypotension-associated adverse events (IHAAE) will be compared at baseline and after intervention, using questionnaires. Participants will undergo a 4-week run-in period to assess baseline incidence. The incidence of IHAAE will be calculated by dividing the number of dialysis treatments with one or more symptoms attributable to IHAAE as a percentage of the total number of dialysis treatments with a completed questionnaire.
  After randomization and the intervention, the occurence of IHAAE will be measured in both arms for another four weeks.
  Differences in incidence of IHAAE between groups will be analyzed using ANCOVA, adjusting for baseline IHAAE, pre-dialysis blood pressure and the use of anti-hypertensive agents.
  IHAAE is defined as a systolic blood pressure < 90 mmHg Either symptomatic or asymptomatic, or solely symptoms associated to (impeding) hypotension like dizziness, lightheadedness, sweating, cramps or visuel disturbances.

SECONDARY OUTCOMES:
Baseline incidence of intradialytic hypotension associated adverse events (IHAAE) in the entire study population. | baseline
  Eligible participants will undergo a 4-week run-in period to assess baseline incidence of IHAAE, using questionnaires.
  The incidence of IHAAE will be calculated by dividing the number of dialysis treatments with one or more symptoms attributable to IHAAE as a percentage of by the total number of dialysis treatments with a completed questionnaire.
Reproducibility of absolute blood volume measurement | 2 weeks
  Absolute blood volume (ABV) will be measured twice in the entire study population, at the start of two mid-weekly hemodialysis treatments.
  We will investigate the correlation between these two test results, using Bland Altman Analysis.
Correlation of absolute blood volume measurement with other diagnostic tests to determine blood volume | 2 weeks
  We will calculate antropomorphic blood volume in the whole study population, using the Nadler's formula.
  We will randomly select 10 participants for ABV measurement with the reference method.This technique is based on the isotope-dilution principal using I-251 radiolabeled human serum albumin. Adverse events due to the infusion of radioactive labelled albumin are very rare (0.01-0.1%, <0.01 % anaphylactic reactions). For a 70kg-patient the dose will be 0,02 millisievert. This falls within risk category I according to the International Commission on Radiological Protection (ICRP). This is the lowest risk category with a statistical probability of less than five in a million to develop radiation induced cancer. Annual background radiation level in the Netherlands is about 2,5 mSv.
  We will correlate the results of these diagnostic tests to our ABV measurement, using Bland Altman analysis.
Sensitivity, specificity | 10 weeks
  We will use the values of absolute volume measurement and incidence of IHAAE to calculate sensitivity, specificity of the previously defined critical threshold of normalized blood volume of 65 ml/kg for the occurrence of IHAAE.
positive predictive value, negative predictive value | 10 weeks
  We will use the values of absolute volume measurement and incidence of IHAAE to calculate positive and negative predictive value of the previously defined critical threshold of normalized blood volume of 65 ml/kg for the occurrence of IHAAE.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Jean Vleming, dr, Principal Investigator — HagaZiekenhuis
Locations (1):
- HagaZiekenhuis, The Hague, Netherlands

IPD SHARING:
Plan to Share IPD: No